CLINICAL TRIAL: NCT06064734
Title: Low-Frequency REpetitive TRanscranial Magnetic Stimulation in ACute Ischemic StrokE Within 48 Hours (RETRACE-I): A Randomized, Open-label, Evaluator-blinded, Phase 2 Pilot Trial
Brief Title: Low-Frequency REpetitive TRanscranial Magnetic Stimulation in ACute Ischemic StrokE Within 48 Hours
Acronym: RETRACE-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2023001
Record Dates: First submitted 2023-08-24; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Stroke, Acute; Stroke, Ischemic
Keywords: Acute Ischemic Stroke; LF-rTMS; Phase 2 Pilot Trial
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigators involved in the clinical evaluation of the patients remained blinded to treatment grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LF-rTMS (Experimental): H 4 Coil (stimulation site: prefrontal cortex, insular lobe),1-Hz rTMS, stimulation intensity RMT 100%,1200 pulses/session, two sessions (2400 pulses)/day (interval ≥2 hours), lasting about half an hour each time, the total duration of treatment was 3 days (6 sessions,7200 pulses).
  Interventions: Device: LF-rTMS
- Control (No Intervention): Routine treatment.

INTERVENTIONS:
Device: LF-rTMS — H 4 Coil (stimulation site: prefrontal cortex, insular lobe),1-Hz rTMS, stimulation intensity RMT 100%,1200 pulses/session, two sessions (2400 pulses)/day (interval ≥2 hours), lasting about half an hour each time, the total duration of treatment was 3 days (6 sessions,7200 pulses).
  Arms: LF-rTMS

SUMMARY:
This is a multicenter, open-label, evaluator-blinded, investigator-initiated, randomized clinical trial, to evaluate the clinical efficacy and safety of LF-rTMS in reducing infarct size, reducing disability rate and improving functional outcome in patients with acute ischemic stroke within 48 hours after stroke onset.

DETAILED DESCRIPTION:
The target population of this study was patients with clinically diagnosed AIS who had an acute occlusion of the responsible vessel in the anterior circulation and were not scheduled for intravenous thrombolysis and/or endovascular therapy, the time from stroke onset to the start of study intervention was less than 48-hours.

Enrolled patients were randomly assigned in a 1:1 ratio to either the"LF-rTMS group" or the"Control group" to receive:

1. LF-rTMS group: H 4 Coil (stimulation site: prefrontal cortex, insular lobe),1-Hz rTMS, stimulation intensity RMT 100%,1200 pulses/session, two sessions (2400 pulses)/day (interval ≥2 hours), lasting about half an hour each time, the total duration of treatment was 3 days (6 sessions,7200 pulses).
2. Control group: received routine treatment.

All the above therapeutic interventions were conducted by trained TMS operators. Except for the study intervention, the subjects in both groups received clinical routine diagnosis and treatment which were not affected by the intervention.

All patients were followed up until the 90th day after randomization to evaluate the clinical efficacy and safety of LF-rTMS in reducing infarct size, reducing disability rate and improving functional outcome in patients with acute ischemic stroke within 48 hours after stroke onset.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, gender is not limited;
2. Acute ischemic stroke of anterior circulation was diagnosed clinically
3. mRS 0-1 score before onset;
4. 6 ≤ NIHSS ≤25 at randomization;
5. Within 48 hours of stroke onset;
6. No thrombolysis therapy or thrombectomy is planned;
7. Obtain informed consent signed by the patient himself or by his legal authorized representative.

Exclusion Criteria:

1. TMS contraindications include metallic foreign bodies in the head, pacemaker, implantable drug pumps, cochlear implants, etc.
2. Epilepsy or history of epilepsy, intracranial hypertension, tumor and other serious neurological disorders;
3. Midline displacement and brain parenchymal mass effect seen in head CT and other images;
4. Head CT or MRI showed bilateral acute cerebral infarction and involved insular infarction;
5. Evidence of acute intracranial hemorrhage;
6. A history of congenital or acquired hemorrhagic disease, coagulation factor deficiency, or thrombocytopenia disease;
7. After blood pressure control, the systolic blood pressure was still ≥180 mmHg or the diastolic blood pressure was ≥110 mmHg;
8. Known recent or current serum creatinine exceeding 1.5 times the upper limit of normal or estimated glomerular filtration rate (EGFR) < 60 mL/min;
9. Patients during pregnancy or lactation and within 90 days of planned pregnancy;
10. Patients with severe mental disorders or dementia who can not cooperate with informed consent and follow-up;
11. Patients with malignancy or severe systemic disease and expected survival of less than 90 days;
12. Participants in other clinical intervention studies within 30 days before randomization or who were participating in other clinical intervention studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-28 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Infarct growth | 3 days
  Infarct growth at 3 days was calculated as the absolute difference between the baseline core infarct volume and the 3 days post-randomization infarct volume.
Proportion of Early neurological improvement (ENI) | 3 days
  Proportion of patients with a reduction of ≥4 on the NIHSS, compared with the baseline score or an NIHSS of 0 or 1
Symptomatic intracranial hemorrhage | 3 days
  The proportion of symptomatic intracranial hemorrhage

SECONDARY OUTCOMES:
Final infarct volume | 3 days
  Final infarct volume
△NIHSS score | 3 days
  Change in NIHSS score from baseline
mRS scores of 0-1 | 90 days
  Proportion of patients with mRS scores of 0-1
mRS scores of 0-2 | 90 days
  Proportion of patients with mRS scores of 0-2
Barthel index of ADL | 90 days
  Barthel index of ADL, 0-100 (better)
EQ-5D-5L | 90 days
  The Health Questionnaire (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems."
Montreal Cognitive Assessment (MoCA) total score | 90 days
  Total score of the MoCA Performance on the MoCA (0-30; higher score indicates better performance)
Serious adverse events | 90 days
  The proportion of serious adverse events (SAE)
All-cause deaths | 90 days
  The proportion of all-cause deaths
Symptomatic intracranial hemorrhage | 90 days
  The incidence of symptomatic intracranial hemorrhage
Deterioration of neurological function | 3 days
  The incidence of deterioration of neurological function (NIHSS increase ≥4 points)
Stroke recurrence | 90 days
  Recurrence rate of symptomatic stroke (cerebral infarction, cerebral hemorrhage)
Adverse events (AE) | 90 days
  The proportion of adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tian tan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No